CLINICAL TRIAL: NCT01729403
Title: A Single Centre, Randomized, Double-Blind, Placebo-Controlled, Phase II Study to Assess the Efficacy of Aleglitazar on Insulin Sensitivity in Patients With Type 2 Diabetes Mellitus (T2D) Who Are Inadequately Controlled With Metformin Monotherapy
Brief Title: A Study of The Effect of Aleglitazar on Insulin Sensitivity in Patients With Type 2 Diabetes Mellitus Who Are Inadequately Controlled With Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WC28038
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — aleglitazar; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Aleglitazar (Experimental)
  Interventions: Drug: aleglitazar; Drug: metformin
- Placebo (Placebo Comparator)
  Interventions: Drug: metformin; Drug: placebo

INTERVENTIONS:
Drug: aleglitazar — 150 mcg orally daily, 16 weeks
  Arms: Aleglitazar
Drug: metformin — patients will continue on their existing dose and regimen of metformin (but not more than the maximum dose specified in the label)
Drug: placebo — orally daily, 16 weeks
  Arms: Placebo

SUMMARY:
This single-center, randomized, double-blind, placebo-controlled study will evaluate the effect of aleglitazar on insulin sensitivity in patients with type 2 diabetes mellitus who are inadequately controlled on metformin monotherapy. Patients will be randomized to receive either aleglitazar 150 mcg or placebo orally daily for 16 weeks, in addition to their existing dose and regimen of metformin.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 30 to 70 years of age inclusive at screening
* Type 2 diabetes mellitus patients treated with stable metformin therapy for at least 12 weeks prior to screening; metformin dose should not exceed the maximum dose specified in the label
* HbA1c >/= 6.5% and </= 9% at screening and baseline
* Fasting plasma glucose </= 13.3 mmol/L (</= 240 mg/dl) at screening and baseline
* Body mass index (BMI) >/= 25 at screening; BMI >/= 27 for subjects with HbA1c < 7%
* Stable weight +/- 5% for at least 12 weeks prior to screening

Exclusion Criteria:

* Women who are pregnant, intending to become pregnant during the study period, currently lactating women, or women of child-bearing potential not using highly effective, medically approved birth control methods
* Diagnosis or history of type 1 diabetes mellitus, diabetes resulting from pancreatic injury, or secondary forms of diabetes
* Acute metabolic diabetic complications such as ketoacidosis or hyperosmolar coma within the past 6 months
* Any previous treatment with a thiazolidinedione or with a dual peroxisome proliferator activated receptor (PPAR) agonist
* Any body weight lowering or lipoprotein-modifying therapy (e.g. fibrates) within 12 weeks prior to screening with the exception of stable (>/= 1 month) statin therapy
* History of bariatric surgery or currently undergoing evaluation for bariatric surgery
* Prior intolerance to fibrate
* Treatment with any anti-diabetic medication other than metformin in the last 12 weeks prior to screening and/or herbal/over-the-counter preparations that may affect glycemic control within 12 weeks prior to screening
* Clinically apparent liver disease
* Positive for hepatitis B, hepatitis C or HIV infection
* Clinical evidence of anemia
* Symptomatic congestive heart failure (New York Heart Association Class II-IV) at screening
* Myocardial infarction, acute coronary syndrome, or transient ischemic attack/stroke within 6 months prior to screening
* Known macular edema at screening or prior to screening visit
* Uncontrolled hypertension despite stable (for at least 4 weeks) anti-hypertensive treatment
* Diagnosed and/or treated malignancy (except for treated cases of basal cell skin cancer, in situ carcinoma of the cervix or in situ prostate cancer) within the past 5 years
* Chronic oral or parenteral corticosteroid treatment (> 2 weeks) within 3 months prior to screening
* History of active substance abuse (including alcohol) within the past 2 years or positive test result for drugs of abuse or alcohol prior to first dosing
* Presence of any absolute or relative contraindication for the conduct of magnetic resonance imaging (MRI) investigation

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in whole-body insulin sensitivity as assessed by M-value (Insulin-stimulated glucose disposal rate) | from baseline to Week 16

SECONDARY OUTCOMES:
Change in hepatic insulin sensitivity (basal index of hepatic insulin resistance) | from baseline to Week 16
Change in parameters of beta cell function (first and second phase insulin secretion) | from baseline to Week 16
Change in HbA1c | from baseline to Week 16
Change in lipid profile | from baseline to Week 16
Change in mean 24h blood pressure | from baseline to Week 16
Change in hepatic fat content measured by magnetic resonance spectroscopy (MRI) | from baseline to Week 16
Change in fat content/distribution in the abdominal region measured by MRI | from baseline to Week 16
Change in total body fat content measured by air displacement phlethysmography | from baseline to Week 16
Change in homeostatic indexes of insulin sensitivity assessed by Homeostasis Model Assessment for Insulin Sensitivity (HOMA-IS) | from baseline to Week 16
Change in markers of cardiovascular risk (high sensitivity C-reactive protein, adiponectin, free fatty acid) | from baseline to Week 16
Safety: Incidence of adverse events | 22 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Neuss, Germany